CLINICAL TRIAL: NCT05245305
Title: The Effect of Mindfulness-Based Stress Reduction Program on Mental Status and Care Burden of Psychotic Patients' Families
Brief Title: The Effect of Mindfulness-Based Stress Reduction Program
Acronym: Mindfulness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Munevver Bogahan, Principal Investigator, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: munevverbghn; Münevver Boğahan (Registry Identifier: Münevver Boğahan)
Record Dates: First submitted 2022-01-24; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: MBSR; Caregiver
Keywords: MBSR; Anxiety; Hopelessness; Care burden; Nursing
MeSH Terms: conditions — Anxiety Disorders; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, two-arm randomized controlled clinical trial Masking: Single (Participant)
Who Masked: Participant
Masking Description: 56 caregiver family members who meet the inclusion criteria and agree to participate in the study will be assigned to the experimental and control groups by simple randomization by an independent researcher who is not included in the study. After the assignments, the statistician will put the 56 family members in which group in sealed envelopes and hand them over to the researcher. The researcher and participants will not know the intervention and control groups until they open the envelope at this stage (single blinding).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBSR Intervention (Experimental): The intervention group will take part in mindfulness-based stress reduction (MBSR) program led by a certified MBSR instructor via Zoom. The MBSR program was structured as 11 weeks, taking into account the characteristics of the participants.
  Interventions: Other: Mindfulness Based Stress Reduction Program
- Control (No Intervention): No intervention was applied to the control group. Data will be collected from the control group simultaneously with the study group.

INTERVENTIONS:
Other: Mindfulness Based Stress Reduction Program — The intervention was structured as 11 weeks, taking into account the group. The program takes 2-2.5 hours per week. The program includes raisin exercise, body scanning meditation, breath awareness meditation, sitting meditation, mindfull movement, walking meditation, vision meditation, compassion meditation,mindfulness communication and day of silence.
  Other Names: MBSR
  Arms: MBSR Intervention

SUMMARY:
This randomized controlled study evaluate the effect of the Mindfulness-Based Stress Reduction Program on the state-trait anxiety, hopelessness, self-compassion and care burden of the families of psychotic patients. The hypothesis of this study is that the Mindfulness-Based Stress Reduction Program improves the state-trait anxiety, hopelessness, self-compassion and care burden of the families of psychotic patients.

DETAILED DESCRIPTION:
Introduction: One of the chronic mental diseases, psychosis causes social and economic losses by negatively affecting the patient's feelings, thoughts and behaviors, interpersonal relations, work and social harmony, and the patient and family may experience different difficulties. With the transition to the community-based model in the provision of mental health services, the relatives of the patients have become the primary caregivers in the care of the patient and their responsibilities have increased even more.When the family is considered as a system, there is a constant interaction between the parts of the system and the change in the patient in case of illness can affect the whole family.When the disease occurs, one of the family members has to take care of the sick individual and caregivers experience emotional (decreased self-esteem, restlessness, depression, insomnia, social isolation, etc.), social (restriction of entertaining, relaxing and leisure time activities, reduction in the role of self-care, etc.). ) and economically (expenses not covered by social security creating an additional burden, reducing working hours, etc.). It is emphasized that psychosocial interventions for families increase the perception of social support, self-efficacy and satisfaction with treatment among caregivers, and reduce the perceived burden and recurrence of the disease.However, the high level of emotional expression and perceived stress of the families may trigger the recurrence of the disease. For this reason, family is naturally emphasized as an important factor in the recovery of the individual with a psychotic illness. Therefore, rehabilitation processes should be aimed not only at patients, but also towards caregivers. One of the interventions used for this purpose today is the Mindfulness-Based Stress Reduction (MBSR) program, which is an evidence-based intervention that teaches skills to reduce stress and manage challenging emotions in a group setting. Although the MBSR intervention is usually aimed at people with chronic physical and mental illnesses, the purpose of the intervention is not to replace medical treatment, but can be used as a supplement, supportive, preventive, complementary or simply a stand-alone method to heal patients. In this respect, it is thought that it is important for psychiatric nurses to use the MBSR program, which is a complementary, supportive, preventive and protective program, in the protection and strengthening of mental health in family members who care for psychosis patients. When the literature is examined, it is emphasized that the MBSR program has positive effects on caregiver family members. In this context, this study is planned to determine the effect of the Mindfulness-Based Stress Reduction Program on the state-trait anxiety, hopelessness, self-compassion and care burden of the families of psychotic patients.

Methods: In the study, 60 family members caring for an individual with psychotic illness were randomly assigned to the study and control groups. 11-week MBSR program will be apply to study group (n = 28). No intervention will be made to the control group (n = 28). The primary outcome of the study is the effect of MBSR on the state-trait anxiety, hopelessness, and self-compassion levels of caregiver family members. The secondary outcome of the study is the effect of MBSR on the caregiving burden of family members. Data will be collected pre-intervention, post-intervention, 3 and 6 months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old
* Able to read and understand Turkish
* Taking care of the sick individual at home
* Living in the same house with the sick individual
* No psychiatric illness
* No problems with movement, sight, hearing or understanding
* Volunteer to participate in the study
* Able to access the internet with their phone or computer
* Those who did not receive any other psychological therapy during their working dates
* No previous meditation experience
* Having no practice in daily mind-body practices

Exclusion Criteria:

* Under 18 years old
* Can't read and understand Turkish
* Any psychiatric illness receiving another psychological therapy on working dates
* Meditation experience before the study; having practice in daily mind-body practices
* Having problems with movement, vision, hearing, understanding
* Not willing to participate in the study
* Participants who participated in more than 50% of a mindfulness-based intervention prior to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-05-15 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Anxiety will be evaluated using the State-Trait Anxiety Scale | Change from preintervention, on average 1 week upon completion of the intervention, 3 months and 6 months after the intervention.
  The total score obtained from both scales varies between 20 and 80. It states that 0-19 points mean no anxiety, 20-39 points mean mild, 40-59 points mean moderate, 60-79 points mean severe anxiety, and individuals with a score of 60 and above need professional help.

SECONDARY OUTCOMES:
Care burden will be assessed using the Caregiver Burden Scale. | Change from preintervention, on average 1 week upon completion of the intervention, 3 months and 6 months after the intervention.
  A score between 22 and 110 is taken from the scale. Obtained points; It is evaluated by grading as "light load" between 22-46, "medium load" between 47-55, "severe load" between 56-110.
Hopelessness will be measured using the Beck Hopelessness Scale. | Change from preintervention, on average 1 week upon completion of the intervention, 3 months and 6 months after the intervention.
  The score range of the scale is 0-20. When the scores obtained are high, hopelessness in the individual is considered high
Self-compassion will be assessed using the Self-Compassion Scale. | Change from preintervention, on average 1 week upon completion of the intervention, 3 months and 6 months after the intervention.
  To calculate the total self-compassion score, the "self-judgmental", "social isolation" and "over-identification" subscale items are reverse coded.
  Then, the self-compassion level is calculated by taking the average of all the items.
  The higher the score for each sub-dimension, the higher the level of self-compassion.
Focus Group Interview Questionnaire I | Within 1 week postintervention
  Focus Group Interview Questionnaire I was created by the researcher in order to evaluate the experiences of the individuals in the study group regarding the MBSR program. There are five questions in the form.

CONTACTS AND LOCATIONS:
Overall Officials: Münevver Boğahan, Assistant, Principal Investigator — Mersin University
Locations (1):
- Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caqueo-Urizar A, Miranda-Castillo C, Lemos Giraldez S, Lee Maturana SL, Ramirez Perez M, Mascayano Tapia F. An updated review on burden on caregivers of schizophrenia patients. Psicothema. 2014 May;26(2):235-43. doi: 10.7334/psicothema2013.86. PMID 24755026
- [Background] Liu Z, Chen QL, Sun YY. Mindfulness training for psychological stress in family caregivers of persons with dementia: a systematic review and meta-analysis of randomized controlled trials. Clin Interv Aging. 2017 Sep 22;12:1521-1529. doi: 10.2147/CIA.S146213. eCollection 2017. PMID 29026290
- [Background] Smith JM, Bright KS, Mader J, Smith J, Afzal AR, Patterson C, Dimitropolous G, Crowder R. A pilot of a mindfulness based stress reduction intervention for female caregivers of youth who are experiencing substance use disorders. Addict Behav. 2020 Apr;103:106223. doi: 10.1016/j.addbeh.2019.106223. Epub 2019 Nov 30. PMID 31838440
- [Background] Stjernsward S, Hansson L. Outcome of a web-based mindfulness intervention for families living with mental illness - A feasibility study. Inform Health Soc Care. 2017 Jan;42(1):97-108. doi: 10.1080/17538157.2016.1177533. Epub 2016 May 31. PMID 27245198
- [Background] Williams H, Simmons LA, Tanabe P. Mindfulness-Based Stress Reduction in Advanced Nursing Practice: A Nonpharmacologic Approach to Health Promotion, Chronic Disease Management, and Symptom Control. J Holist Nurs. 2015 Sep;33(3):247-59. doi: 10.1177/0898010115569349. Epub 2015 Feb 11. PMID 25673578
- [Background] Whitebird RR, Kreitzer M, Crain AL, Lewis BA, Hanson LR, Enstad CJ. Mindfulness-based stress reduction for family caregivers: a randomized controlled trial. Gerontologist. 2013 Aug;53(4):676-86. doi: 10.1093/geront/gns126. Epub 2012 Oct 15. PMID 23070934
- [Derived] Bogahan M, Yilmaz S, Yilmaz M. Effects of Mindfulness-Based Stress Reduction Program on the Mental Health and Care Burden in Family Caregivers of Individuals with Psychosis. Community Ment Health J. 2025 Oct 17. doi: 10.1007/s10597-025-01527-z. Online ahead of print. PMID 41105316
- See also: An updated review on burden on caregivers of schizophrenia patients — https://pubmed.ncbi.nlm.nih.gov/24755026/
- See also: Mindfulness training for psychological stress in family caregivers of persons with dementia: a systematic review and meta-analysis of randomized controlled trials — https://pubmed.ncbi.nlm.nih.gov/29026290/
- See also: A pilot of a mindfulness based stress reduction intervention for female caregivers of youth who are experiencing substance use disorders — https://pubmed.ncbi.nlm.nih.gov/31838440/
- See also: Outcome of a web-based mindfulness intervention for families living with mental illness - A feasibility study — https://pubmed.ncbi.nlm.nih.gov/27245198/
- See also: Mindfulness-Based Stress Reduction in Advanced Nursing Practice: A Nonpharmacologic Approach to Health Promotion, Chronic Disease Management, and Symptom Control — https://pubmed.ncbi.nlm.nih.gov/25673578/
- See also: Mindfulness-based stress reduction for family caregivers: a randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/23070934/